CLINICAL TRIAL: NCT00072410
Title: Single-Dose, Cohort Study of Increasing Doses of Yttrium-90 Conjugated to Humanized Monoclonal Antibody 3S193 (90Y-hu3S193) in Patients With Advanced Ovarian Cancer
Brief Title: Radiolabeled Monoclonal Antibody in Treating Patients With Advanced Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000339682; MSKCC-03069 (Other: Memorial Sloan-Kettering Cancer Center); LUD2001-018 (Other: Ludwig Institute for Cancer Research)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer; stage III ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — 90Y-CHX-A''-DTPA-hu3S193; Yttrium-90

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Patients received a single intraperitoneal (IP) dose of 10 mg of hu3S193 radiolabeled with 10 millicuries (mCi) 90Y and 5mCi 111In-hu3S193 to enable imaging after dosing.
  Interventions: Biological: 90Y-hu3S193; Biological: 111In-hu3S193
- Cohort 2 (Experimental): Patients received a single intraperitoneal (IP) dose of 10 mg of hu3S193 radiolabeled with 15 millicuries (mCi) 90Y and 5mCi 111In-hu3S193 to enable imaging after dosing.
  Interventions: Biological: 90Y-hu3S193; Biological: 111In-hu3S193

INTERVENTIONS:
Biological: 90Y-hu3S193 — Patients received a single dose of 10 mg of hu3S193 radiolabeled with the intended dose (mCi) of 90Y.
  Other Names: humanized monoclonal antibody 3S193 radiolabeled with 90Y
Biological: 111In-hu3S193 — Patients received a single dose of 5 mCi 111In-hu3S193 together with the 90Y-hu3S193.
  Other Names: humanized monoclonal antibody 3S193 radiolabeled with 111In

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and deliver radioactive tumor-killing substances to them without harming normal cells. Giving radiolabeled monoclonal antibody directly into the abdominal cavity may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of giving radiolabeled monoclonal antibody therapy directly into the abdominal cavity in treating patients who have advanced ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and maximum tolerated dose of intraperitoneally (IP) administered yttrium-90 (90Y) radiolabeled monoclonal antibody (mAB) hu3S193 (90Y-hu3S193) in patients with advanced ovarian epithelial cancer.

Secondary

* Determine the localization and whole body and abdominal clearance of 90Y-hu3S193 using indium-111 (111In) radiolabeled hu3S193 and gamma camera imaging.
* Determine the serum pharmacokinetics of hu3S193 using gamma well counting.
* Determine the antibody response as measured by human anti-human antibody response (HAHA).

OUTLINE: This is a dose-escalation study of the yttrium-90 radiolabeled monoclonal antibody, 90Y-hu3S193.

Patients received technetium (99mTc-sulfur colloid) IP and underwent abdominal imaging on day 1. Provided the distribution of the 99mTC-sulfur colloid was deemed adequate, patients then received 90Y-hu3S193 IP. 111In-hu3S193 was also administered IP over 30 minutes on day 1 to enable gamma camera imaging. Within 3-5 hours after antibody administration, patients underwent whole body imaging and single-photon emission-computed tomography (SPECT) imaging of the abdomen and pelvis.

Cohorts of 3-6 patients were to receive escalating doses of 90Y-hu3S193 until the maximum tolerated dose (MTD) was determined. The MTD was defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients were to be followed every 3 months for at least 2 years and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria

1. Histologically confirmed non-mucinous ovarian adenocarcinoma.
2. Persistent or recurrent intraperitoneal cancer following platinum/taxane-based therapy for Stage 3 ovarian cancer.
3. Patients with residual disease < 2cm will be candidates for this study.
4. The following laboratory and clinical results within the last 2 weeks prior to study day 1:

   Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; Platelet count ≥ 100 x 10^9/L; Serum bilirubin ≤ 2.0 mg/dL; Aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN); Alanine aminotransferase (ALT) ≤ 2.5 x ULN; Serum creatinine ≤2.0 mg/dL; Forced expiratory volume (FEV1) ≥60% of predicted; Forced vital capacity (FVC) ≥60% of predicted; Diffusion capacity ≥55% of predicted; Left ventricular ejection fraction (LVEF) ≥50%;
5. Karnofsky performance status ≥ 70.
6. Before any trial-specific procedures or treatment can be performed, the patient or legally authorized guardian or representative must give witnessed written informed consent for participation in the trial.
7. Placement of an intra-abdominal catheter at the time of surgery.

Exclusion Criteria

1. Active parenchymal disease (i.e., Stage IV International Federation of Gynecology and Obstetrics (FIGO) classification).
2. Presence of symptomatic extra abdominal metastases.
3. Known central nervous system (CNS) tumor involvement.
4. Clinically significant heart disease (New York Heart Association Class III or IV).
5. ECG demonstrating clinically significant arrhythmias or evidence of prior myocardial infarction.
6. Other serious illnesses, eg, serious infections requiring antibiotics, bleeding disorders that may limit the amount of antibody they can tolerate or render them ineligible for surgery.
7. Chronic inflammatory bowel disease.
8. Chemotherapy, biologic therapy, or immunotherapy within 4 weeks prior to enrollment.
9. Pregnancy or lactation.
10. Patients who are positive for human anti-human antibodies (HAHA) and/or who have received a murine monoclonal antibody.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2003-11 (Actual); Primary Completion 2005-05 (Actual); Study Completion 2006-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaitanya R. Divgi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Patients received a single intraperitoneal (IP) dose of 10 mg of hu3S193 radiolabeled with 10 millicuries (mCi) 90Y and 5 mCi 111In-hu3S193 to enable imaging after dosing.
  90Y-hu3S193: Patients received a single dose of 10 mg of hu3S193 radiolabeled with the intended dose (mCi) of 90Y.
  111In-hu3S193: Patients received a single dose of 5 mCi 111In-hu3S193 together with the 90Y-hu3S193.
- Cohort 2: Patients received a single intraperitoneal (IP) dose of 10 mg of hu3S193 radiolabeled with 15 millicuries (mCi) 90Y and 5 mCi 111In-hu3S193 to enable imaging after dosing.
  90Y-hu3S193: Patients received a single dose of 10 mg of hu3S193 radiolabeled with the intended dose (mCi) of 90Y.
  111In-hu3S193: Patients received a single dose of 5 mCi 111In-hu3S193 together with the 90Y-hu3S193.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 3 | 4
Completed | 3 | 1
Not Completed | 0 | 3
Not completed — Progressive disease | 0 | 3

BASELINE CHARACTERISTICS:
Population: All patients who entered the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose-limiting Toxicities (DLTs)
Description: All adverse events were graded according to the National Cancer Institute Common Toxicity Criteria (CTC) Scale (Version 2.0, published April 30, 1999). DLT was defined as:
  * Any Grade 3 or greater non-hematological toxicity (except for alopecia, nausea, and vomiting, defined separately below)
  * Any Grade alopecia
  * Grade 4 nausea or vomiting ≥ 5 days duration.
  * Any Grade 4 hematological toxicity (except for toxicity of ≤ 5 days duration without growth factor, platelet, or transfusion support). To be dose limiting, an adverse event must be definitely, probably, or possibly related to the administration of the investigational agent.
Time Frame: Up to day 56
Population: All patients who entered the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

2. Secondary Outcome: Clearance as Measured by the Half-life (T1/2) of the Elimination Phase
Description: Serum samples were taken 5 min, 1 hour, and 2 hours after end of infusion, twice on study day 2, and daily on study days 3 to 7, 8, 15 and 22. Serum samples were analyzed in a gamma well counter. Elimination half-life (T1/2) was generated by fitting effective clearance to a monoexponential curve.
Time Frame: Up to 22 days
Population: All patients who entered the study and had serum samples taken at the specified times. Patient No. 5 in Cohort 2 did not have Day 22 blood drawn and was not included in the mean value.
Measure: Mean (Full Range); unit: days
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 3
days | 2.43 [2.31 to 2.57] | 2.28 [2.22 to 2.34]

3. Secondary Outcome: Number of Patients With Human Anti-human Antibodies (HAHA) After Treatment
Description: Blood samples were taken at baseline and on days15, 28 and 56. HAHA was measured by BIACORE.
Time Frame: Up to day 56
Population: All patients who entered the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 56 days
Description: All adverse events occurring during the study were recorded on the patient's case report form. Adverse events were graded according to the National Cancer Institute Common Toxicity Criteria (CTC) Scale (Version 2.0, published April 30, 1999).
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/3 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=4)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Dizziness (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No